CLINICAL TRIAL: NCT01360320
Title: Minimizing the Risk of Metachronous Adenomas of the Colorectum With Green Tea Extract -MIRACLE-
Acronym: MIRACLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: University of Ulm (Other); KKS Netzwerk (Network); Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Thomas Seufferlein, Prof. Dr. med., Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MIRACLE
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Serrated Adenomas; Colorectal Tubular Adenomas; Colorectal Villous Adenomas; Colorectal Tubulovillous Adenomas
Keywords: Green tea; polyphenol; catechin; EGCG; Epigallocatechin gallate; colorectal adenoma; adenoma prevention; colon cancer prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Green tea extract (Experimental): Powdered decaffeinated green tea extract of Camellia Sinensis, packed in hard gelatine capsules containing either 150 mg EGCG, bid for 3 years
  Interventions: Dietary Supplement: Green tea extract of Camellia Sinensis
- Placebo (Placebo Comparator): Placebo, packed in hard gelatine capsules, bid for 3 years
  Interventions: Dietary Supplement: Green tea extract of Camellia Sinensis followed by placebo

INTERVENTIONS:
Dietary Supplement: Green tea extract of Camellia Sinensis — Powdered decaffeinated green tea extract of Camellia Sinensis, packed in hard gelatine capsules containing either 150 mg EGCG
  * Run-in period with 150mg EGCG two times daily (p.o) for 4 weeks
  * 150mg EGCG two times daily (p.o.) over the course of three years.
  * Colonoscopy after 3 years
  Arms: Green tea extract
Dietary Supplement: Green tea extract of Camellia Sinensis followed by placebo — Powdered decaffeinated green tea extract of Camellia Sinensis, packed in hard gelatine capsules containing either 150 mg EGCG
  * Run-in period with 150mg EGCG two times daily (p.o.) for 4 weeks
  * Placebo two times daily (p.o.) over the course of three years
  * Colonoscopy after 3 years
  Arms: Placebo

SUMMARY:
This is a randomized, placebo controlled, multicentric trial to investigate the effect of diet supplementation with green tea extract containing 300mg epigallocatechin gallate (EGCG), the major polyphenol of green tea, on the recurrence of colon adenomas.

DETAILED DESCRIPTION:
Prevention of colorectal cancer is a major health care issue because of the high incidence of this cancer. So far, pharmaceutical chemoprevention has not gained widespread acceptance due to side effects of the chemopreventive agents used. Nutraceuticals such as polyphenols from tea plants have demonstrated remarkable therapeutic and preventive effects in molecular, epidemiological and clinical trials. However, controlled trials demonstrating the efficacy of nutraceuticals fo the prevention of colorectal cancer are largely missing.

The investigators present this randomized, placebo controlled, multicentric trial to investigate the effect of diet supplementation with green tea extract containing 300mg epigallocatechin gallate (EGCG), the major polyphenol of green tea, on the recurrence of colon adenomas.

Patients who underwent polypectomy for colonic polyps will be randomized after a one month verum run-in period to receive either 150mg EGCG two times daily or placebo over the course of three years. The beneficial safety profile of decaffeinated green tea extract, the quantifiable and known active content EGCG, and the accumulating evidence on its cancer preventive potential require in our view a validation of this compound for the "nutriprevention" of colorectal adenoma. Good accessibility and low costs might render this nutraceutical a top candidate for a wider use as food supplement in colon cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

* Between 50-80 years of age
* Histologically confirmed colorectal adenomas or serrated lesions removed during colonoscopy within the last 6 months
* Good performance status (ECOG < 2) at study entrance
* Written informed consent.

Exclusion Criteria:

* History of hereditary nonpolyposis colorectal cancer (HNPCC) or familial adenomatous polyposis (FAP)
* History of colon or rectal cancer, other concomitant cancers with the exemption of basalioma or curative treated cancers without actual anticancer medication.
* Intestinal malabsorption, short bowel syndrome or surgical bowel interventions leading to malabsorption
* Liver failure (hepatitis, cirrhosis, elevation of liver enzymes ALT, AST or bilirubin to more than 2.5 fold of the reference levels)
* Inflammatory bowel disease
* Regular intake of NSAIDs (also Cox2 inhibitors) for more than 3 months per year except of low-dose aspirin (100 mg per day)
* Immunosuppressive medication
* Impaired capacity to consent or who are impaired in swallowing a pill
* Regular consumption of green tea extract as nutritional supplement (with a content of EGCG of more than 100mg per day) of longer than 6 months during the past two years
* Allergic reactions towards green tea

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Incidence of metachronous colorectal adenomas (tubulovillous, tubular, villous and serrated lesions) at the 3 year follow-up colonoscopy | 3 years

SECONDARY OUTCOMES:
Occurrences of colorectal adenomas or mucosal lesions | 3 years
Number of colorectal adenomas or mucosal lesions | 3 years
Size of colorectal adenomas or mucosal lesions | 3 years
Localization of colorectal adenomas or mucosal lesions | 3 years
Histological subtypes of colorectal adenomas or mucosal lesions | 3 years
Invasive growth of colorectal adenomas or mucosal lesions | 3 years
Incidence of colorectal carcinoma | 3 years
Translational research | 3 years
  Genetic and biochemical biomarkers for recurrence of adenoma or development of dysplasia and carcinoma (blood samples and histological in tissue samples of the colorectal lesions)
Toxicity and feasibility | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Julia Stingl, Prof.Dr.med, Study Chair — Federal Institute for Drugs and Medical Devices, Bonn, Germany; Thomas Seufferlein, Prof.Dr.med., Principal Investigator — University Hospital Ulm, Ulm, Germany
Locations (21):
- Germany (21):
  - Ostalb-Klinikum Aalen, Medizinische Klinik 1, Sekretariat Prof. Kleber, Aalen
  - Klinikum Altenburger Land, Gastroenterologie, Altenburg
  - Klinikum Augsburg, III. Med. Klinik, Augsburg
  - Krankenhaus Bietigheim-Bissingen, Klinik für Innere Medizin, Gastroenterologie, Hämato-Onkologie, Bietigheim-Bissingen
  - Krankenhaus Buchholz, Abteilung Innere Medizin, Buchholz
  - Kliniken der Stadt Köln gGmbH, Krankenhaus Holweide -Medizinische Klinik-, Cologne
  - Klinikum Esslingen, Klinik für Innere Medizin, Onkologie, Gastroenterologie, Esslingen am Neckar
  - Universitätsklinikum der Ernst-Moritz-Arndt-Universität Greifswald, Klinik und Poliklinik für Innere Medizin A, Greifswald
  - Dr. Zeisler, Praxis für Innere Medizin und Gastroenterologie, Halle
  - Dres. Fechner/Behrens/Steudel - Gastroenterologisch-Onkologische Praxisklinik, Halle
  - Dr. Frank-Gleich Praxis für Innere Medizin und Gastroenterologie, Halle
  - Universitätsklinikum Halle, Klinik für Innere Medizin I, Halle
  - Klinikum Ludwigsburg, Medizinische Klinik I, Ludwigsburg
  - Diakoniekrankenhaus Mannheim, Medizinische Klinik II, Mannheim
  - II. Medizinische Klinik und Poliklinik der TU München, Klinikum rechts der Isar, Munich
  - Klinik Mühldorf Abt.Gastroenterologie, Mühldorf
  - Klinikum Bogenhausen, Interdisziplinäre Onkologische Tagklinik, München
  - Regio Kliniken Pinneberg, Pinneberg
  - Klinikum St. Elisabeth, I. Medizinische Klinik, Straubing
  - Universitätsklinikum Ulm, Klinik für Innere Medizin I, Ulm
  - Evangelisches Krankenhaus Wesel, Abteilung Innere Medizin, Wesel

REFERENCES:
- [Background] Stingl JC, Ettrich T, Muche R, Wiedom M, Brockmoller J, Seeringer A, Seufferlein T. Protocol for minimizing the risk of metachronous adenomas of the colorectum with green tea extract (MIRACLE): a randomised controlled trial of green tea extract versus placebo for nutriprevention of metachronous colon adenomas in the elderly population. BMC Cancer. 2011 Aug 18;11:360. doi: 10.1186/1471-2407-11-360. PMID 21851602
- [Derived] Melzer A, Sturm N, Rohlmann F, Muche R, Stingl J, Ettrich TJ, Seufferlein T. Interest in complementary and alternative medicine among participants in a study on cancer prevention by green tea extract - results from an expert-based survey of MIRACLE trial participants. BMC Complement Med Ther. 2025 Oct 2;25(1):350. doi: 10.1186/s12906-025-05087-3. PMID 41039315
- [Derived] Seufferlein T, Ettrich TJ, Menzler S, Messmann H, Kleber G, Zipprich A, Frank-Gleich S, Algul H, Metter K, Odemar F, Heuer T, Hugle U, Behrens R, Berger AW, Scholl C, Schneider KL, Perkhofer L, Rohlmann F, Muche R, Stingl JC. Green Tea Extract to Prevent Colorectal Adenomas, Results of a Randomized, Placebo-Controlled Clinical Trial. Am J Gastroenterol. 2022 Jun 1;117(6):884-894. doi: 10.14309/ajg.0000000000001706. Epub 2022 Feb 25. PMID 35213393
- [Derived] Scholl C, Lepper A, Lehr T, Hanke N, Schneider KL, Brockmoller J, Seufferlein T, Stingl JC. Population nutrikinetics of green tea extract. PLoS One. 2018 Feb 21;13(2):e0193074. doi: 10.1371/journal.pone.0193074. eCollection 2018. PMID 29466429
- See also: Related Info — http://www.gruenteestudie.de
- See also: Related Info — http://www.krebshilfe.de